CLINICAL TRIAL: NCT05445518
Title: Jump Start Plus: Coronavirus Disease (COVID-19) Support to Improve Resiliency and Mitigate Risks in Childcare Centers Serving Children From Low-income Ethnic Minority Backgrounds.
Brief Title: Jump Start Plus COVID-19 Support
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ruby Natale, Associate Professor of Clinical Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20220115; R01HD105474 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jump Start Plus COVID Support (JS+CS) Group (Experimental): Participants in this group will receive the Jump Start Plus COVID Support intervention for 24 months.
  Interventions: Behavioral: Jump Start Plus COVID Support
- Healthy Caregivers-Healthy Children (HC2) Control Group (Active Comparator): Participants in this group will receive the Healthy Caregivers-Healthy Children intervention for 24 months.
  Interventions: Behavioral: Healthy Caregivers-Healthy Children (HC2)

INTERVENTIONS:
Behavioral: Jump Start Plus COVID Support — The Jump Start Plus COVID Support intervention is a resiliency program that provides behavior management and safety programs administered weekly via zoom.
  Arms: Jump Start Plus COVID Support (JS+CS) Group
Behavioral: Healthy Caregivers-Healthy Children (HC2) — The HC2 intervention is an obesity prevention program that provides nutrition and healthy activities programs administered weekly via Zoom.
  Arms: Healthy Caregivers-Healthy Children (HC2) Control Group

SUMMARY:
The purpose of the study is to further develop and examine the Jump Start Plus COVID Support (JS+CS) program, which encourages improved psychosocial functioning by promoting resiliency in childcare centers.

ELIGIBILITY:
Center Inclusion Criteria:

1. Have greater than 30 children ages 2- to 5-years old
2. Serve low-income families
3. Reflect the ethnic diversity of Miami-Dade County (60%Hispanic, 20% Non-Hispanic Black, 20% Non-Hispanic White

Child Inclusion Criteria:

1. Child ages 2-5 years old
2. Child enrolled in a childcare center

Exclusion Criteria:

* Children with feeding tubes or those that bring their own meals.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Health Environment Rating Scale Scores | Baseline, Up to 3 years
  The Health Environment Rating Scale has a total score ranging from 0 to 70 with higher scores indicating healthier practices
Change in Strengths and Difficulties Questionnaire Scores | Baseline, Up to 3 years
  The Strengths and Difficulties Questionnaire is a total difficulties score that ranges from 0 to 40 with higher scores indicating less child behavior concerns.
Change in Devereux Early Childhood Assessments Scores | Baseline, Up to 3 years
  The Devereux Early Childhood Assessments is a measure with a range of score from 0 to 100 with higher score on Behavior Concerns indicating more problem behaviors and a lower score on Initiative, Self-Control, Attachment indicated better protective factors.

SECONDARY OUTCOMES:
Change in Brief Resilient Coping Scale Scores | Baseline, Up to 3 years
  The Brief Resilient Coping Scale is a measure with a range of score from 4 to 20 with a higher score indicating better coping.
Change in Childcare Worker Job Stress Index Scores | Baseline, Up to 3 years
  The Childcare Worker Job Stress Index is a total score that ranges from 22 to 110 with higher scores indicating higher levels of stress
Change in Every Day Stressors Index Scores | Baseline, Up to 3 years
  The Every Day Stressors Index is a total score that ranges from 0 to 80 with higher scores indicating higher levels of stress.
Change in Healthy Caregivers-Healthy Children Survey | Baseline, Up to 3 years
  Teacher and parents complete this survey on the number of reported nutrition and physical activity practices
Change in Teacher Opinion Survey | Baseline, up to 3 years
  The Teacher Opinion survey is a measure with a range of score from 12 to 44 with higher score indicating better self-efficacy as it relates to teaching practices.

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Natale, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No